CLINICAL TRIAL: NCT01730924
Title: A Randomised Study Comparing Pulmonary Vein Isolation Using SmartTouch® Catheter With or Without Real-time Contact Force Data. The SMART Trial
Brief Title: Comparison of Pulmonary Vein Isolation Using SmartTouch® Catheter With or Without Real-time Contact Force Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Prof Richard Schilling, Professor of Cardiology, Queen Mary University of London
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 008205 QM
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Ablation; Pulmonary Vein Isolation
Keywords: Atrial fibrillation; Contact force; Ablation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (2):
- Contact force available (Other)
  Interventions: Procedure: Pulmonary vein isolation using contact force sensing catheter
- Contact force not available (Other)
  Interventions: Procedure: Pulmonary vein isolation using contact force sensing catheter

INTERVENTIONS:
Procedure: Pulmonary vein isolation using contact force sensing catheter

SUMMARY:
The most widely used approach for the invasive treatment of paroxysmal atrial fibrillation is catheter ablation, by which radiofrequency energy is used to heat the tip of an ablation catheter to deliver targeted burns on the inner surface of the heart. The aim of this approach is to cause electrical isolation of the pulmonary veins. The purpose of this study is to evaluate whether the information which can be derived from the latest catheter technologies - on the degree of contact force between the catheter and the heart - affects the time to perform the procedure, or the outcomes as a result of it. Patients undergoing pulmonary vein isolation will be randomised to having their procedure performed with the contact force information available to the operator, or not available. The time taken to achieve pulmonary vein isolation is the primary end-point of the study.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years, Symptomatic paroxysmal atrial fibrillation (defined as ECG proven episodes of atrial fibrillation which are self limiting and last less than 7 days on each occasion)

Exclusion Criteria:

Inability or unwillingness to receive oral anticoagulation Previous ablation procedure for atrial fibrillation Unwillingness or inability to complete the required follow up arrangements Persistent atrial fibrillation Prior prosthetic mitral valve replacement or severe structural cardiac abnormality Known severe left ventricular systolic function (ejection fraction <35%) Known hypertrophic or infiltrative cardiomyopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to achieve pulmonary vein isolation in patients undergoing catheter ablation for paroxysmal atrial fibrillaiton

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, London, United Kingdom

REFERENCES:
- [Derived] Ullah W, McLean A, Tayebjee MH, Gupta D, Ginks MR, Haywood GA, O'Neill M, Lambiase PD, Earley MJ, Schilling RJ; UK Multicentre Trials Group**. Randomized trial comparing pulmonary vein isolation using the SmartTouch catheter with or without real-time contact force data. Heart Rhythm. 2016 Sep;13(9):1761-7. doi: 10.1016/j.hrthm.2016.05.011. Epub 2016 May 9. PMID 27173976